CLINICAL TRIAL: NCT05621772
Title: MARS-PD: Meridian Activation Remedy System for Parkinson's Disease - A Single-center, Rater-blinded, Parallel Randomized Controlled Trial
Brief Title: Meridian Activation Remedy System for Parkinson's Disease
Acronym: MARS-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, HoRyong Yoo, Prof. Dr., Daejeon University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DJ_PD_21_02
Record Dates: First submitted 2022-11-04; First posted 2022-11-18 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A Single-center, Rater-blinded, Parallel Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Meridian Activation Remedy System for Parkinson's Disease) (Experimental): Meridian Activation Remedy System for Parkinson's Disease (MARS-PD) treatment (16 times/8 weeks total, 2 times/week)
  Interventions: Other: Meridian Activation Remedy System for Parkinson's Disease (MARS-PD)
- Control group (Usual Care) (No Intervention): Usual care (all participants will be allowed to continue their prescribed medication and treatment (except Korean Medicine therapy), and they will not receive any additional treatment or therapy in the research institute), and lifestyle advice (all participants will receive a smart band and application-based guidance about their lifestyle)

INTERVENTIONS:
Other: Meridian Activation Remedy System for Parkinson's Disease (MARS-PD) — MARS-PD is a complex therapy developed by researchers to enhance the synergistic effects of acupuncture and exercise.
  Arms: Experimental group (Meridian Activation Remedy System for Parkinson's Disease)

SUMMARY:
In this study, the investigators aim to evaluate the clinical efficacy and cost-effectiveness of MARS-PD. Conventional, usual care will be used as the comparator because this trial aims to assess the add-on effect of MARS-PD. The investigators hypothesize that the complex therapy will relieve motor and nonmotor symptoms, improve gait performance, and enhance neuroplasticity in PD patients, and will be safe and cost-effective.

DETAILED DESCRIPTION:
This study is a randomized controlled trial conducted at a single center with raters blinded to the intervention. We will look at the clinical effect of MARS-PD, consisting of 16 interventions over an 8-week period, in 88 individuals with Parkinson's disease. Patients will be assigned to either the experimental (n=44) or control (n=44) groups at random. he experimental group will receive the MARS intervention, while the control group will receive usual care only. The treatment duration is 8 weeks, followed by a 12-week follow-up. The primary outcome is the change in MDS-UPDRS Part III (Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III) score from baseline to 8 weeks. Secondary outcomes include assessments such as MDS-UPDRS, International Physical Activity Questionnaire Short Form, Parkinson Self Questionnaire, Parkinson's Disease Sleep Scale, Timed Up and Go test, GAITRite metrics, Functional Near-Infrared Spectroscopy measurements, smart band results, gut microbiome composition and diversity, and iris connective tissue texture.

ELIGIBILITY:
Inclusion Criteria:

1. 45 to 75 years of age
2. Patients with PD, diagnosed according to the United Kingdom Parkinson's Diseases Society Brain Bank Criteria
3. Hoehn and Yahr scale stage I to III
4. Patients who have voluntarily decided to participate in the clinical study and signed the informed consent form

Exclusion Criteria:

1. Clinically unstable patients (e.g., elevated aspartate transaminase (AST) or alanine aminotransferase (ALT) more than three-fold the upper limit of normal in the research institute's laboratory, heart failure, respiratory failure, etc.)
2. Patients who are planning to undergo deep brain stimulation within the study period
3. Pregnant or lactating women
4. Patients with MMSE-K (Mini-Mental State Exam) score of 18 or less
5. If there has been a change in the dosage of antiparkinsonian drugs (e.g., L-dopa, COMT (catechol-O-methyltransferase) inhibitor, Dopamine agonist, MAO-B (monoamine oxidase B) inhibitor, etc.) according to a doctor's prescription within the last 4 weeks prior to enrollment
6. Patients who are receiving manual therapy, exercise therapy, or rehabilitation therapy for Parkinson's disease according to a doctor's prescription within the last 4 weeks prior to enrollment, or are planning to receive such therapy within the study period
7. Patients who are not suitable for participation in this clinical study according to the judgment of the researcher

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale Part Ⅲ | Change from baseline MDS-UPDRS Part Ⅲ score at 8 weeks
  MDS-UPDRS Part Ⅲ (maximum: 132, minimum: 0; higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale Part Ⅲ | Change from baseline MDS-UPDRS Part Ⅲ score at 4 and 12 weeks
  MDS-UPDRS Part Ⅲ
International Physical Activity Questionnaire Short Form | Change from baseline IPAQ score at 4, 8 and 12 weeks
  IPAQ
Parkinson Self Questionnaire | Change from baseline Parkinson Self Questionnaire results at 4, 8 and 12 weeks
  Parkinson Self Questionnaire, developed by researchers
Parkinson's disease Sleep Scale | Change from baseline PDSS score at 4, 8 and 12 weeks
  PDSS
Timed up and go test | Change from baseline TUG time in seconds at 8 and 12 weeks
  TUG
GAITRite Electronic Walkway Platinum | Change from baseline GAITRite parameters at 8 and 12 weeks
  GAITRite
Functional near-infrared spectroscopy | Change from baseline fNIRS results at 8 and 12 weeks
  fNIRS
Smart band outcomes | Change from baseline daily steps at 4, 8 and 12 weeks
  Number of steps per day
Iris imaging 1 | Iris connective tissue texture, baseline
  Visible light image
Iris imaging 2 | Iris connective tissue density, baseline
  Infrared image
Movement Disorder Society Unified Parkinson's Disease Rating Scale | Change from baseline MDS-UPDRS score at 4, 8 and 12 weeks
  MDS-UPDRS
Gut microbiome test | Change from baseline gut microbiome analysis results at 8 weeks
  Gut microbiome diversity and composition, fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Ho Ryong Yoo, Prof. Dr., Principal Investigator — Daejeon University
Locations (1):
- Clinical Trial Center, Daejeon Korean Medicine Hospital of Daejeon University, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hur WJ, Seo JW, Park MS, Yoo HR. Visual self-reporting for symptom communication in Parkinson's disease. Technol Health Care. 2026 Feb 5:9287329251414326. doi: 10.1177/09287329251414326. Online ahead of print. PMID 41641966
- [Derived] Park MS, Park S, Kang JY, Jung IC, Yoo H. The efficacy and safety of MARS-PD: Meridian activation remedy system for Parkinson's disease-A single-center, assessor and statistician-blinded, parallel-group randomized, controlled trial protocol. PLoS One. 2024 May 6;19(5):e0303156. doi: 10.1371/journal.pone.0303156. eCollection 2024. PMID 38709746